CLINICAL TRIAL: NCT05248399
Title: Vale+ Tu Salud: Corner-Based Randomized Trial to Test a Latino Day Laborer Program Adapted to Prevent COVID-19.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Maria Eugenia Fernandez-Esquer, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-20-1389 (Rapid phase); 1R01MD016328-01 (NIH)
Record Dates: First submitted 2022-02-17; First posted 2022-02-21 (Actual); Results first posted 2023-07-20 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-06

CONDITIONS: COVID-19
Keywords: Latino Day Laborers
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Cluster Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID-19 Group Problem Solving plus Standard of Care (Experimental)
  Interventions: Behavioral: COVID-19 Group Problem Solving; Behavioral: Standard of Care
- Standard of Care (Active Comparator)
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: COVID-19 Group Problem Solving — The COVID-19 Group Problem Solving component incorporates popular education activities aimed at: developing social cohesion among LDLs; building awareness about COVID-19 risks and protective behaviors; and developing a plan of action to reduce theirs and their peers' risk for COVID-19 transmission. The intervention will be developed to take place over a ~30-45-minute period in order to fit within the corner context of LDLs waiting for employment, and will be delivered by promoters from our team and the community partner agency, Fe & Justicia Workers Center. Following the completion of the intervention, a health promoter will be trained as a navigator assist participants who wish to get vaccinated by providing them with information about near-by vaccination sites that they can visit to get vaccinated. If needed, the promotor will assist them with making their vaccine appointment.
  Arms: COVID-19 Group Problem Solving plus Standard of Care
Behavioral: Standard of Care — The standard of care consists of the distribution of brochures containing COVID-19 prevention information.

SUMMARY:
The purpose of this study is to adapt and pilot test the feasibility of implementing a corner-based risk reduction program that aims to assist Latino day laborers (LDL) in their efforts to adhere to COVID-19 mitigation practices, including receiving the COVID-19 vaccine, using personal protective equipment (PPE), and practicing social distancing.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Hispanic or Latino
* Be present at the corner for the purposes of looking for work

Exclusion Criteria:

* Have not been previously hired to work at a corner
* Symptoms of COVID-19 in the previous 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria E Fernandez-Esquer, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Constantin AM, Noertjojo K, Sommer I, Pizarro AB, Persad E, Durao S, Nussbaumer-Streit B, McElvenny DM, Rhodes S, Martin C, Sampson O, Jorgensen KJ, Bruschettini M. Workplace interventions to reduce the risk of SARS-CoV-2 infection outside of healthcare settings. Cochrane Database Syst Rev. 2024 Apr 10;4(4):CD015112. doi: 10.1002/14651858.CD015112.pub3. PMID 38597249

RESULTS

PARTICIPANT FLOW:
Groups:
- COVID-19 Group Problem Solving Plus Standard of Care: The COVID-19 Group Problem Solving component incorporates popular education activities aimed at: developing social cohesion among LDLs; building awareness about COVID-19 risks and protective behaviors; and developing a plan of action to reduce theirs and their peers' risk for COVID-19 transmission. The intervention will be developed to take place over a ~30-45-minute period in order to fit within the corner context of LDLs waiting for employment, and will be delivered by promoters from our team and the community partner agency, Fe & Justicia Workers Center. Following the completion of the intervention, a health promoter will be trained as a navigator assist participants who wish to get vaccinated by providing them with information about near-by vaccination sites that they can visit to get vaccinated. If needed, the promotor will assist them with making their vaccine appointment.
  The Group Problem Solving arm will also receive standard of care, which consists of the distribution of brochures containing COVID-19 prevention information.
- Standard of Care: The Control arm will receive standard of care, which consists of the distribution of brochures containing COVID-19 prevention information.
Period: Overall Study
Arm/Group | COVID-19 Group Problem Solving Plus Standard of Care | Standard of Care
Started | 101 | 99
Completed | 84 | 82
Not Completed | 17 | 17

BASELINE CHARACTERISTICS:
Population: One of the participants who started the study and who received the Group Problem Solving intervention was found to not be a day laborer, and so that participant was excluded and their data are not included in the baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | COVID-19 Group Problem Solving Plus Standard of Care | Standard of Care | Total
Number analyzed (Participants) | 100 | 99 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age data were not collected for 3 in the Group Problem Solving plus Standard of Care arm and for 1 in the Standard of Care arm.
  years
    number analyzed (Participants) | 97 | 98 | 195
    (all) | 49.4 (11.3) | 44.0 (12.6) | 46.7 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 99 | 99 | 198
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 100 | 99 | 199
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 100 | 99 | 199
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 100 | 99 | 199

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Change in COVID-19 Vaccination Status Assessed by a Survey
Time Frame: Baseline, 4 weeks post intervention
Population: Baseline and 4 week data were only collected for 81 in the COVID-19 Group Problem Solving plus Standard of Care arm and for 80 in the Standard of Care arm.
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Group Problem Solving Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 81 | 80
Participants
  Number of participants not vaccinated at baseline and who did not receive vaccine after baseline | 24 | 36
  Number of participants not vaccinated at baseline and who received vaccine after baseline | 1 | 0
  Number of participants vaccinated at baseline and did not receive a repeat vaccine after baseline | 49 | 36
  Number of participants vaccinated at baseline and who received a repeat vaccine after baseline | 7 | 8

2. Secondary Outcome: Change in Mask Wearing Frequency as Assessed by Change in Mean Mask Use Total Score on a Survey
Description: Participants were asked seven items measuring how often they had worn a mask in different situations (e.g. while at the corner) in the last 30 days (baseline) or since their baseline survey (one month post test). Responses were recorded as 1 = Never; 2 = Sometimes; 3 = Many Times; 4 = All the Time. Participants could refuse to answer any item or respond that the particular item did not apply to them (for example., they do not wear a mask on public transport because they do not take public transport) . These responses were treated as missing.
  Mask Use score was computed as the mean score of the items with a non-missing response, and mean mask use total score could range from 1 to 4. Change in mean mask use score is reported, and change score was computed by subtracting the baseline score from the post test score, with a negative change score indicating a decrease in mask use.
Time Frame: Baseline, 4 weeks post intervention
Population: Baseline and 4 week data were only collected for 84 in the COVID-19 Group Problem Solving plus Standard of Care arm and for 82 in the Standard of Care arm.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | COVID-19 Group Problem Solving Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 84 | 82
scores on a scale | -0.38 (0.95) | -0.32 (0.80)

3. Secondary Outcome: Change in Social Distancing as Assessed by Change in Mean Social Distancing Total Score on a Survey
Description: Participants were asked six items measuring how often they had practiced Social Distancing in different situations (e.g. while at the worksite) in the last 30 days (baseline) or since their baseline survey (one month post test). Responses were recorded as 1 = Never; 2 = Sometimes; 3 = Many Times; 4 = All the Time. Participants could refuse to answer any item or respond that the particular item did not apply to them. These responses were treated as missing
  Social Distancing score was computed as the mean score of the items with a non-missing response, and mean mask use total score could range from 1 to 4. Change in mean mask use score is reported and was computed by subtracting the baseline score from the post test score, with a negative change score indicating a decrease in social distancing.
Time Frame: Baseline, 4 weeks post intervention
Population: Baseline and 4 week data were only collected for 83 in the COVID-19 Group Problem Solving plus Standard of Care arm and for 82 in the Standard of Care arm.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | COVID-19 Group Problem Solving Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 83 | 82
scores on a scale | -0.13 (0.86) | -0.09 (0.82)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | COVID-19 Group Problem Solving Plus Standard of Care | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/99
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/99
Other Adverse Events (participants affected / at risk) | 0/101 | 0/99

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/99/NCT05248399/Prot_SAP_000.pdf